CLINICAL TRIAL: NCT03476967
Title: Effect of Panretinal Photocoagulation on Confocal Laser Scanning Ophthalmoscopy and Stereo Photographic Parameters of the Optic Disc Topography in Diabetic Retinopathy Patients
Brief Title: Effect of Laser Treatment for Diabetic Retinopathy on the Optic Disc Topography
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Other Study IDs: USaoPauloGH 12423
Record Dates: First submitted 2018-03-09; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Diabetic Retinopathy
Keywords: optic disc topography; panretinal photocoagulation; confocal scanning laser ophthalmoscopy; stereoscopic disc photographs; diabetic retinopathy; optic nerve head parameters
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pretreatment x Posttreatment: The group was evaluated through non-invasive complementary examinations before laser therapy and at the 1-year follow-up visit to analyze possible optical disc alterations that may occur after retinal panretinal photocoagulation in patients with proliferative diabetic retinopathy.
  Interventions: Procedure: Panretinal photocoagulation

INTERVENTIONS:
Procedure: Panretinal photocoagulation — In cases of proliferative diabetic retinopathy (PDR), panretinal photocoagulation (PRP) is the first-line treatment. Although PRP reduces the risk of severe vision loss, it has been shown that laser energy can cause destruction to all layers of retina including the ganglion cells and the retinal nerve fiber layer (RNFL), and therefore generate visual field defects similar to that observed in glaucomatous damage. In such cases, visual field testing can be less helpful to evaluate glaucomatous damage in PDR patients treated with PRP.

SUMMARY:
This study analyzed diabetic patients without evidence of glaucoma who underwent panretinal photocoagulation to determine the effect on optic disc topographic parameters in non-glaucomatous patients with proliferative diabetic retinopathy (PDR).

DETAILED DESCRIPTION:
Glaucoma and proliferative diabetic retinopathy (PDR) are two very prevalent diseases that often coexist. Previous literature suggest that panretinal photocoagulation may somehow lead to optic disk cupping. Therefore, evaluation of the optic disc cupping and of possible glaucomatous damage in patients with diabetic retinopathy can be difficult, especially after PRP treatment. The purpose of this study is to determine the long-term effect of PRP on optic disc topographic parameters in non-glaucomatous patients with PDR using Heidelberg retina tomograph (HRT) parameters and stereo photography. The Investigators found that PRP does not cause morphological optic disk changes in diabetic PDR patients after one year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PDR (due to type 1 or 2 diabetes mellitus)
* intraocular pressure < 18 mmHg
* nonglaucomatous optic disc characteristics at fundus examination
* vertical cup-to-disc (C/D) ratio <0.7
* absence of media opacities

Exclusion Criteria:

* previous diagnosis of glaucoma
* family history of glaucoma
* neuroophthalmic disease
* uveitis
* retinal artery or vein occlusion
* optic disc neovascularization
* diabetic macular edema (DME)
* corneal opacity
* previous laser photocoagulation treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients followed in the ophthalmology department of Hospital das Clínicas da FMUSP who have type I or II diabetes mellitus and present severe or very severe non proliferative diabetic retinopathy or proliferative diabetic retinopathy in cases where retinal panphotocoagulation is indicated.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Cup area | 12 months
  Change in cup area (mm2) measured by Heidelberg retinal tomograph (HRT) before and one year after PRP

CONTACTS AND LOCATIONS:
Overall Officials: Leandro Zacharias, Study Director — Division of Ophthalmology, University of São Paulo Medical School, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months after study publication
Access Criteria: Data access request will be reviewed by study director. Requestors will be required to sign a Data access agreement